CLINICAL TRIAL: NCT00510679
Title: A Randomized Controlled Trial of Post-Training Supports for Health Workers Trained in the Use of Integrated Management of Childhood Illness Guidelines in Ouémé Department, Benin
Brief Title: Study of Post-Training Supports for Health Workers in Benin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Benin (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDC-NCID-3279
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-08

CONDITIONS: Malaria; Pneumonia; Diarrhea; Measles; Malnutrition
Keywords: Benin; child health; developing country; health services research; health worker performance; Integrated Management of Childhood Illness
MeSH Terms: conditions — Malaria; Pneumonia; Diarrhea; Measles; Malnutrition | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Health worker supports (supervision, job aids, incentives)

SUMMARY:
The objective of this study was to determine the effectiveness and cost-effectiveness of a package of interventions to support health workers in Benin (in West Africa) who had been trained to use Integrated Management of Childhood Illness guidelines (i.e., guidelines intended to improve the treatment of childhood illnesses).

DETAILED DESCRIPTION:
Integrated Management of Childhood Illness (IMCI) is a child health strategy in developing countries with a goal of improving the treatment of illnesses at first-level health facilities through the use of clinical practice guidelines. The World Health Organization (WHO) recommends implementing the guidelines with an 11-day training course. There is a concern that health workers might not master all aspects of the guidelines and that health worker performance may deteriorate over time. In 1999, Benin (in West Africa) was planning to implement IMCI. In response to concerns about how well health workers would follow IMCI guidelines, interventions were designed to support health workers after IMCI training: 1) regular supervision of health workers; 2) supervision of supervisors; 3) job aids; and 4) non-financial incentives for health workers. These interventions were intended to be used together. The objective of this study was to determine the effectiveness and cost-effectiveness of the package of interventions to support IMCI-trained health workers in Benin.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for health facilities were: 1) public and licensed private health facilities providing outpatient services, and 2) the level of care was appropriate for use of Integrated Management of Childhood Illness (IMCI) guidelines.
* Inclusion criteria for consultations were children 1 week - 59 months old seen for any illness during regular working hours (typically 8am-6pm) on weekdays.

Exclusion Criteria:

* Health facilities in which the level of care was not appropriate for use of Integrated Management of Childhood Illness (IMCI) guidelines(i.e., one referral hospital and one sub-specialty hospital).

Ages: 1 Week to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1577 (Actual)
Dates: Start 1999-07; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Proportion of children with potentially life-threatening illnesses who received recommended treatment, according to Integrated Management of Childhood Illness guidelines. | 3 years
Proportion of children with potentially life-threatening illnesses who received recommended treatment, according to Integrated Management of Childhood Illness guidelines, or adequate treatment. | 3 years
Mean proportion of needed case management tasks that were performed during consultations. | 3 years

SECONDARY OUTCOMES:
Proportion of children with pneumonia who received recommended treatment, according to Integrated Management of Childhood Illness guidelines. | 3 years
Proportion of children with malaria who received recommended treatment, according to Integrated Management of Childhood Illness guidelines. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rowe K Alexander, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- All eligible health facilities, Entire Department of Oueme and Plateau, Oueme and Plateau, Benin

REFERENCES:
- [Background] Rowe AK, Onikpo F, Lama M, Deming MS. Risk and protective factors for two types of error in the treatment of children with fever at outpatient health facilities in Benin. Int J Epidemiol. 2003 Apr;32(2):296-303. doi: 10.1093/ije/dyg063. PMID 12714553
- [Background] Rowe AK, Lama M, Onikpo F, Deming MS. Design effects and intraclass correlation coefficients from a health facility cluster survey in Benin. Int J Qual Health Care. 2002 Dec;14(6):521-3. doi: 10.1093/intqhc/14.6.521. No abstract available. PMID 12515339
- [Background] Rowe AK, Lama M, Onikpo F, Deming MS. Health worker perceptions of how being observed influences their practices during consultations with ill children. Trop Doct. 2002 Jul;32(3):166-7. doi: 10.1177/004947550203200317. No abstract available. PMID 12139161
- [Background] Rowe AK, Onikpo F, Lama M, Cokou F, Deming MS. Management of childhood illness at health facilities in Benin: problems and their causes. Am J Public Health. 2001 Oct;91(10):1625-35. doi: 10.2105/ajph.91.10.1625. PMID 11574325
- [Derived] Rowe AK, Onikpo F, Lama M, Deming MS. Evaluating health worker performance in Benin using the simulated client method with real children. Implement Sci. 2012 Oct 8;7:95. doi: 10.1186/1748-5908-7-95. PMID 23043671
- [Derived] Rowe AK, Onikpo F, Lama M, Deming MS. The rise and fall of supervision in a project designed to strengthen supervision of Integrated Management of Childhood Illness in Benin. Health Policy Plan. 2010 Mar;25(2):125-34. doi: 10.1093/heapol/czp054. Epub 2009 Nov 18. PMID 19923206
- [Derived] Osterholt DM, Onikpo F, Lama M, Deming MS, Rowe AK. Improving pneumonia case-management in Benin: a randomized trial of a multi-faceted intervention to support health worker adherence to Integrated Management of Childhood Illness guidelines. Hum Resour Health. 2009 Aug 27;7:77. doi: 10.1186/1478-4491-7-77. PMID 19712484